CLINICAL TRIAL: NCT01419483
Title: A Phase I Trial of a Ketogenic Diet With Concurrent Chemoradiation for Pancreatic Cancer.
Brief Title: Ketogenic Diet With Concurrent Chemoradiation for Pancreatic Cancer
Acronym: KETOPAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor accrual
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Nutricia North America (Industry)
Responsible Party: Principal Investigator, Bryan Allen, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201102772; 1R21CA161182 (NIH)
Record Dates: First submitted 2011-07-28; First posted 2011-08-18 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic neoplasms; Pancreatic cancer; Ketogenic Diet; radiotherapy; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketogenic diet (Experimental): Diet designed to maintain elevated ketone levels during therapy
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — A ketogenic diet matching the fat to carbohydrate + proteins in Keto-Cal(R) 4:1 by Nutricia North America.

SUMMARY:
This study investigates if using a very low carbohydrate diet during combined chemotherapy and radiation therapy is safe and if it can be tolerated by patients.

DETAILED DESCRIPTION:
Standard treatment for pancreatic cancer includes chemotherapy concurrent with radiation therapy (chemoradiation).

This study is a phase I trial to determine the safety of dietary manipulation during chemoradiation for pancreatic cancer. Specifically, pre-clinical data from mouse studies indicates a ketogenic diet increases tumor cell killing.

Participants will:

* Utilize a specialized ketogenic diet designed by bionutritional services of the clinical research unit. This diet begins 2 days before chemoradiation and continues through at least 5 weeks of chemoradiation.
* Have blood drawn for research purposes weekly to determine measurements of oxidative stress
* Have urine collected sporadically through the study to determine measurements of oxidative stress
* Keep a diary of concomitant medications, side effects, and blood sugars
* Have follow-up to monitor for outcomes and overall survival

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cytological or histological diagnosis of adenocarcinoma arising in the pancreas. Adenosquamous cancers will be acceptable.
* Cancer should be staged via AJCC as IIA, IIB, or III (T3 or T4, any N, M0)
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky > 50%, see Appendix A).
* Hypertensive medication should be initiated or increased for optimal blood pressure control according to standard public health guidelines prior to starting the ketogenic diet.
* Patients must have normal organ and marrow function as defined below:
* leukocytes ≥ 3,000/mm3
* absolute neutrophil count ≥ 1,500/mm3
* platelets ≥ 100,000/mm3
* total bilirubin < 3.0 mg/dl
* Hgb A1C < or = to 8%
* AST(SGOT) < or = 5 X institutional upper limit of normal OR a stable or a decreasing test value in patients who have undergone placement of an intrabiliary stent. Both the treating radiation oncologist and medical oncologist must agree that the potential subject's test value is acceptable for study accrual.
* creatinine < 1.5 X institutional upper limit of normal OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Not pregnant. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior abdominal radiotherapy.
* Prior therapy, with the intent to treat, the current diagnosis of pancreatic cancer.
* Known G6PD (glucose-6-phosphate dehydrogenase) deficiency.
* Patients on corticosteroids for any reason.
* Living alone at time of diet initiation.
* Other investigational agents/therapy with the intention to treat the disease under study (observational or imaging trials are acceptable).
* Uncontrolled diabetes defined as a hemoglobin A1C level > 8% (therapeutic action is indicated at greater than 8%).
* Diabetes mellitus is not exclusionary provided the patient is not maintained with either oral medications or insulin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations, or any other condition that would limit compliance with study requirements as determined by study team members.
* Pregnant or lactating women: The risks of radiation and chemotherapy to a fetus are well documented.

Female and male patients of all ethnic groups will be eligible for treatment in these protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (Safety) | Weekly for 8 weeks
  Categorize and quantify adverse events in subjects implementing a ketogenic diet while undergoing definitive chemoradiation therapy.

SECONDARY OUTCOMES:
Ketone levels | Daily during treatment for 6 weeks
  Quantify blood ketone levels via both finger-stick prior to daily radiation therapy and weekly lab analysis while on a ketogenic diet. Radiation is administered Monday through Friday only.
Blood glucose levels | Daily during treatment for 6 weeks
  Quantify blood glucose levels via finger-stick prior to daily radiation therapy while on a ketogenic diet. Radiation therapy is administered Monday through Friday only.
Oxidative stress parameters | Weeks 1, 2, 3, 4, 5, and 6 of treatment and at 1 month follow-up
  Determine oxidative stress parameters in plasma and urine samples during the course of treatment.
Progression Free Survival (months) | Every 12 months for 60 months
  From date of treatment until the first date of documented progression or date of death, whichever comes first, assessed no less than every 12 months for the first 60 months post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan G. Allen, MD, PhD, Principal Investigator — The Department of Radiation Oncology, The University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

REFERENCES:
- [Result] Zahra A, Fath MA, Opat E, Mapuskar KA, Bhatia SK, Ma DC, Rodman SN III, Snyders TP, Chenard CA, Eichenberger-Gilmore JM, Bodeker KL, Ahmann L, Smith BJ, Vollstedt SA, Brown HA, Hejleh TA, Clamon GH, Berg DJ, Szweda LI, Spitz DR, Buatti JM, Allen BG. Consuming a Ketogenic Diet while Receiving Radiation and Chemotherapy for Locally Advanced Lung Cancer and Pancreatic Cancer: The University of Iowa Experience of Two Phase 1 Clinical Trials. Radiat Res. 2017 Jun;187(6):743-754. doi: 10.1667/RR14668.1. Epub 2017 Apr 24. PMID 28437190